CLINICAL TRIAL: NCT05594329
Title: A Randomized Controlled Trial to Investigate the Neurological, Inflammatory and Metabolic Effects of Acute Mushroom Intervention in Older Adults (OYSACO)
Brief Title: Neurological, Inflammatory and Metabolic Effects of Acute Mushroom Intervention in Older Adults
Acronym: OYSACO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Mushroom Council (Other)
Responsible Party: Principal Investigator, Prof Claire Williams, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 22/10
Record Dates: First submitted 2022-10-11; First posted 2022-10-26 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Cognitive Change; Mood; Metabolism; Inflammatory Response; Satiety
Keywords: Cognition; Mood; Inflammation; Metabolism
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental meal 1 (Experimental): Instant noodle soup containing 2 servings of dried Pleurotus oyster mushroom.
  Interventions: Other: Instant noodle soup containing containing the equivalent of 2 servings (18.78g) of powdered Pleurotus oyster mushroom.
- Experimental meal 2 (Experimental): Instant noodle soup containing 1 serving of dried Pleurotus oyster mushroom.
  Interventions: Other: Instant noodle soup containing containing the equivalent of 1 serving (9.39g) of powdered Pleurotus oyster mushroom.
- Experimental meal 3 (Experimental): Instant noodle soup containing 0.5 serving of dried Pleurotus oyster mushroom.
  Interventions: Other: Instant noodle soup containing containing the equivalent of 0.5 serving (4.70g) of powdered Pleurotus oyster mushroom.
- Control meal (Placebo Comparator): Instant noodle soup containing cornflour and maltodextrin in a 2.5:1 ratio.
  Interventions: Other: Control instant noodle soup

INTERVENTIONS:
Other: Instant noodle soup containing containing the equivalent of 2 servings (18.78g) of powdered Pleurotus oyster mushroom. — Ingredients: celery, garlic, ginger, gluten, polyphosphate, parsley, pepper, potassium carbonates, dried Pleurotus oyster mushroom, salt, sodium, sunflower oil, turmeric, yeast extract and wheat flour.
  Arms: Experimental meal 1
Other: Instant noodle soup containing containing the equivalent of 1 serving (9.39g) of powdered Pleurotus oyster mushroom. — Ingredients: cornflour, celery, garlic, ginger, gluten, polyphosphate, parsley, pepper, potassium carbonates, dried Pleurotus oyster mushroom, maltodextrin, salt, sodium, sunflower oil, turmeric, yeast extract and wheat flour.
  Arms: Experimental meal 2
Other: Instant noodle soup containing containing the equivalent of 0.5 serving (4.70g) of powdered Pleurotus oyster mushroom. — Ingredients: cornflour, celery, garlic, ginger, gluten, polyphosphate, parsley, pepper, potassium carbonates, dried Pleurotus oyster mushroom, maltodextrin, salt, sodium, sunflower oil, turmeric, yeast extract and wheat flour.
  Arms: Experimental meal 3
Other: Control instant noodle soup — Ingredients: cornflour, celery, garlic, ginger, gluten, polyphosphate, parsley, pepper, potassium carbonates, maltodextrin, salt, sodium, sunflower oil, turmeric, yeast extract and wheat flour.
  Arms: Control meal

SUMMARY:
This randomized crossover trial (RCT) investigates the acute effect (over a 6-hour period) of a meal containing varying serving sizes (doses) of freeze-dried oyster mushroom powder, on the cognitive behaviour and markers of metabolism and inflammation related to neuronal health in healthy adults aged 60-80 years old. The study will involve a screening visit and four testing visits, with a week interval between each. During the four testing visits, cognitive-mood battery tests will be taken at baseline and then at 2-, 4- and 6-hour intervals following the consumption of the intervention meal. Also, a blood draw will be taken at the end of each testing visit day to allow the determination of inflammatory, metabolic and neuronal markers.

DETAILED DESCRIPTION:
The Pleurotus oyster species is a common edible mushroom rich in ergothioneine, a bioactive compound with known neurocognitive benefits. The aim of the OYSACO RCT is to provide a clearer understanding of how a meal containing varying serving sizes (doses) of freeze-dried oyster mushroom powder, may acutely regulate cognitive improvements in humans during the immediate postprandial period. The investigators will investigate the neurological and physiological changes underlying these benefits.

During the OYSACO RCT, participants will attend the University of Reading, Psychology department on five separate occasions, with a week interval between each visit. Specifically, in the pre-screening phase, to check for eligibility, the participants interested in our study will be sent a link to REDCap containing online versions of a Health and Lifestyle Questionnaire containing basic demographic questions (eg age, sex, heigh, weight, nationality, disease history and medication use) and the Epic Norfolk Food Frequency Questionnaire (FFQ), to assess their habitual dietary intake. Then, participants, will be contacted to attend a 2-hour screening session at our department, during which the participant's weight, height and blood pressure will be checked, along with a finger-prick, to ensure that the participants are not anaemic. Three drops of blood will be taken from the tip of the either the index or ring finger for this measure. Furthermore, participants will complete the Raven's Progressive Matrices (RPM) measure of fluid intelligence and will perform the cognitive battery tasks twice to control for practice effects in the run up to the test session days.

One week after the screening visit, each participant will attend a further four test sessions, each separated by a week, where they will receive a different dose of freeze-dried oyster mushrooms. The order of intervention will be randomised, and participants will be asked to follow a low fibre and flavonoid diet for 48 hours in advance of testing. Before each test visit, the participants will be asked to fast for 12-hours and then to consume only a slice of toast with butter and 1 glass of water at 07:00 a.m., before attending the university. As soon as the participants arrive at our laboratory at 08:00 a.m., baseline cognitive and mood tests will be completed. After completing the baseline measures, the participants will receive one of the 3 mushroom interventions or the control intervention. The procedure on each test day will be identical except for the intervention meal. Specifically, the intervention meals will consist of a noodle soup containing the equivalent of 0.5, 1 and 2 servings of powdered Pleurotus oyster mushroom or a calorie-matched control non-mushroom noodle soup containing a mixture of maltodextrin and cornflour. The ingredients present in the intervention meals are all standard ingredients used in the food industry and are included at safe levels. Allergy information will be available on request. The dried oyster mushroom powder was prepared according to the Federal Good Manufacturing Practices and US Food Guidelines and is certified free from unauthorised pesticides, and microbiological and other contaminants.

Two-hours after consuming the intervention, the participants will be asked to complete the same cognitive and mood tests, and a calorie-matched lunch will then be provided between 12:00-12:30 p.m. containing a chicken sandwich, a packet of crisps and a glass of water. Participants will then be asked to complete the cognitive and mood tests a further two times (4-hours and 6-hours post-intervention) and a blood test will be drawn at the end of the visit.

In addition to the cognitive tests, palatability measures will be taken immediately after the consumption of the intervention meal while at the end of each cognitive test session (at baseline, 2-, 4- and 6-hours), ratings of subjective appetite and fullness will be recorded using an online analogue scale. At the end of the 5-week study, participants will be asked to complete a brief dietary questionnaire, consisting of specialised questions, relating to their habitual mushroom intake.

In terms of cognitive testing, there will be four cognitive task battery sessions taking place at baseline and then at 2-, 4-and 6-hours post-intervention, to assess participants' episodic and working memory, psychomotor and executive function and mood domains. Each battery will be matched for difficulty and order of presentation will be randomised. Although the exact cognitive battery is yet to be confirmed, all tasks will be completed on the computer and should take no longer than 45 minutes to complete. The battery is likely to contain the following or similar tasks:

* Positive and Negative Affect Schedule (PANAS-SF)- In this mood task, participants are asked to rate their emotion on a 5-point Likert scale, in response to 20 mood related adjectives (10 relating to positive emotions and 10 to negative emotions).
* Rey Auditory Verbal Learning Task (RAVLT)- This episodic memory task consists of 5 consecutive free recalls of the same 15 nouns presented as an auditory list (list A), followed by recall of a further 15 nouns presented as an interference list (list B) which is recalled only once. List A is subsequently recalled straight after list B and then again after a longer delay of around 30 minutes.
* Corsi block tapping task (CBTT)- In this spatial working memory task, participants are shown with 9 arranged blocks positioned on a computer screen and are asked to reproduce given sequence by clicking on the blocks (using the mouse) in the same sequence as they see them.
* Simple and complex finger tapping task- In this motor function task, participants tap on a key as quickly as possible with the index finger of their dominant hand for 1 minute. They then tap out a specific sequence using 4 fingers, again for 1 minute.
* Task Switching Task (TST) - In this executive function task, participants view 8 spaced radii of a circle above and below a bold line and a stimulus digit selected from 1-9 (except 5) appears clockwise in each segment, either above or below the bold line. Depending on the stimulus position in the segments, participants perform different tasks with each being switched in every 4 trials.
* RAVLT word recall- After a period of time, participants are asked to recall as many words as possible from list A.
* RAVLT word recognition- In this delayed memory task, participants are shown a sequential list of 50 nouns containing the words from lists A and B from the previously described RAVLT task plus 20 additional words not previously heard, and are asked to indicate those from list A.

During each test day, participants will have one 9-millilitre blood draw taken from their arm, 6-hours after receiving the intervention meal. Following each draw, the serum will be separated via centrifuge and stored at at -80°C until analysis is complete. Whole blood samples will not be stored at any point during the study. Blood serum will be analysed for anti-inflammatory and metabolic ability by measuring the levels of fasting glucose and lipids in the blood, the markers of inflammation, as well as the levels of the brain derived neurotrophic factor (BDNF), a signalling protein known to be related to neuronal signalling and memory function.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 60-80 years old
* Have normal vision and hearing
* Have healthy status
* Have a BMI<30

Exclusion Criteria:

* Smokers or those consuming more than the recommended units of alcohol per week
* Vegetarians/ Vegans
* Being diagnosed with any psychiatric or neurologic conditions (e.g. schizophrenia, depression, cognitive dementia)
* Being diagnosed with cardiometabolic disease (including type II diabetes and cardiovascular disease), or suffer from hypertension or thrombosis related disorders
* Being anaemic
* Currently taking regular vitamin supplements or disease medication such as anticoagulant or antiplatelet medication and antidepressants etc
* Diagnosed with an eating disorder
* Be allergic to mushrooms, or any other nutrients present in the intervention meals

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Change in Positive and Negative Affect Schedule (PANAS-SF) performance | 2-hours post-intervention
  In this validated self-reported mood task, participants are asked to rate their emotion. The PANAS comprises of two distinct affective states (positive and negative), as well as 11 individual affective states (fear, guilt, sadness, surprise, hostility, shyness, joviality, self-assurance, attentiveness, fatigue and serenity). Subjects use a likert scale from 1 - 5 to indicate how the word relates to how they are currently feeling. As this analysis is exploratory all affective states will be explored.
Change in Positive and Negative Affect Schedule (PANAS-SF) performance | 4-hours post-intervention
  In this validated self-reported mood task, participants are asked to rate their emotion. The PANAS comprises of two distinct affective states (positive and negative), as well as 11 individual affective states (fear, guilt, sadness, surprise, hostility, shyness, joviality, self-assurance, attentiveness, fatigue and serenity). Subjects use a likert scale from 1 - 5 to indicate how the word relates to how they are currently feeling. As this analysis is exploratory all affective states will be explored.
Change in Positive and Negative Affect Schedule (PANAS-SF) performance | 6-hours post-intervention
  In this validated self-reported mood task, participants are asked to rate their emotion. The PANAS comprises of two distinct affective states (positive and negative), as well as 11 individual affective states (fear, guilt, sadness, surprise, hostility, shyness, joviality, self-assurance, attentiveness, fatigue and serenity). Subjects use a likert scale from 1 - 5 to indicate how the word relates to how they are currently feeling. As this analysis is exploratory all affective states will be explored.
Change in Immediate Word Recall performance from the Rey Auditory Verbal Learning Task (RAVLT) | 2-hours post-intervention
  This episodic memory task consists of 5 consecutive free recalls of the same 15 nouns presented as an auditory list (list A), followed by recall of a further 15 nouns presented as an interference list (list B) which is recalled only once. List A is subsequently recalled straight after list B and then again after a longer delay of around 30 minutes.
Change in Immediate Word Recall performance from the Rey Auditory Verbal Learning Task (RAVLT) | 4-hours post-intervention
  This episodic memory task consists of 5 consecutive free recalls of the same 15 nouns presented as an auditory list (list A), followed by recall of a further 15 nouns presented as an interference list (list B) which is recalled only once. List A is subsequently recalled straight after list B and then again after a longer delay of around 30 minutes.
Change in Immediate Word Recall performance from the Rey Auditory Verbal Learning Task (RAVLT) | 6-hours post-intervention
  This episodic memory task consists of 5 consecutive free recalls of the same 15 nouns presented as an auditory list (list A), followed by recall of a further 15 nouns presented as an interference list (list B) which is recalled only once. List A is subsequently recalled straight after list B and then again after a longer delay of around 30 minutes.
Change in Corsi Block Tapping Test (CBTT) performance | 2-hours post-intervention
  In this spatial working memory task, participants are shown with 9 arranged blocks positioned on a computer screen and are asked to reproduce a given sequence by clicking on the blocks (using the mouse) in the same sequence as they see them.
Change in Corsi Block Tapping Test (CBTT) performance | 4-hours post-intervention
  In this spatial working memory task, participants are shown with 9 arranged blocks positioned on a computer screen and are asked to reproduce a given sequence by clicking on the blocks (using the mouse) in the same sequence as they see them.
Change in Corsi Block Tapping Test (CBTT) performance | 6-hours post-intervention
  In this spatial working memory task, participants are shown with 9 arranged blocks positioned on a computer screen and are asked to reproduce a given sequence by clicking on the blocks (using the mouse) in the same sequence as they see them.
Change in Simple and complex finger tapping task (SFTT & CFTT) performance | 2-hours post-intervention
  In this motor function task, participants tap on a key as quickly as possible with the index finger of their dominant hand for 1 minute. They then tap out a specific sequence using 4 fingers, again for 1 minute.
Change in Simple and complex finger tapping task (SFTT & CFTT) performance | 4-hours post-intervention
  In this motor function task, participants tap on a key as quickly as possible with the index finger of their dominant hand for 1 minute. They then tap out a specific sequence using 4 fingers, again for 1 minute.
Change in Simple and complex finger tapping task (SFTT & CFTT) performance | 6-hours post-intervention
  In this motor function task, participants tap on a key as quickly as possible with the index finger of their dominant hand for 1 minute. They then tap out a specific sequence using 4 fingers, again for 1 minute.
Change in the Task Switching Task (TST) performance | 2-hours post-intervention
  In this executive function task, participants view 8 spaced radii of a circle above and below a bold line and a stimulus digit selected from 1-9 (except 5) appears clockwise in each segment, either above or below the bold line. Depending on the stimulus position in the segments, participants perform different tasks with each being switched in every 4 trials. A response of higher or lower than 5 is made for trials below the bold line, and even or odd for numbers above the line. Outcome measures include overall accuracy and reaction time (RT) on correct trials, as well as accuracy and RT on trials where there is a 'switch cost' from stimuli moving from below to above the bold line and vice versa.
Change in the Task Switching Task (TST) performance | 4-hours post-intervention
  In this executive function task, participants view 8 spaced radii of a circle above and below a bold line and a stimulus digit selected from 1-9 (except 5) appears clockwise in each segment, either above or below the bold line. Depending on the stimulus position in the segments, participants perform different tasks with each being switched in every 4 trials. A response of higher or lower than 5 is made for trials below the bold line, and even or odd for numbers above the line. Outcome measures include overall accuracy and reaction time (RT) on correct trials, as well as accuracy and RT on trials where there is a 'switch cost' from stimuli moving from below to above the bold line and vice versa.
Change in the Task Switching Task (TST) performance | 6-hours post-intervention
  In this executive function task, participants view 8 spaced radii of a circle above and below a bold line and a stimulus digit selected from 1-9 (except 5) appears clockwise in each segment, either above or below the bold line. Depending on the stimulus position in the segments, participants perform different tasks with each being switched in every 4 trials. A response of higher or lower than 5 is made for trials below the bold line, and even or odd for numbers above the line. Outcome measures include overall accuracy and reaction time (RT) on correct trials, as well as accuracy and RT on trials where there is a 'switch cost' from stimuli moving from below to above the bold line and vice versa.
Change in RAVLT - Delayed Word Recall performance | 2-hours post-intervention
  After a period of time subject are asked to recall as many words as possible from list A.
Change in RAVLT - Delayed Word Recall performance | 4-hours post-intervention
  After a period of time subject are asked to recall as many words as possible from list A.
Change in RAVLT - Delayed Word Recall performance | 6-hours post-intervention
  After a period of time subject are asked to recall as many words as possible from list A.
Change in RAVLT - Word Recognition performance | 2-hours post-intervention
  Following the delayed word recall, words from list A, list B and novel words are displayed sequentially on the screen and participants are asked to indicate which words were from list A only.
Change in RAVLT - Word Recognition performance | 4-hours post-intervention
  Following the delayed word recall, words from list A, list B and novel words are displayed sequentially on the screen and participants are asked to indicate which words were from list A only.
Change in RAVLT - Word Recognition performance | 6-hours post-intervention
  Following the delayed word recall, words from list A, list B and novel words are displayed sequentially on the screen and participants are asked to indicate which words were from list A only.

SECONDARY OUTCOMES:
Visual analogue measure of hunger, satiety, fullness, and prospective food consumption | Baseline
  Satiety Measure recorded on a 100 millimetre scale. Scores closer to 0 millimetres indicate less hunger, less satiety and less fullness - taken as a negative outcome, and less desire for prospective food consumption or consume something sweet, salty, savoury or fatty - taken as a positive outcome.
Visual analogue measure of hunger, satiety, fullness, and prospective food consumption | 2-hours post-intervention
  Satiety Measure recorded on a 100 millimetre scale. Scores closer to 0 millimetres indicate less hunger, less satiety and less fullness - taken as a negative outcome, and less desire for prospective food consumption or consume something sweet, salty, savoury or fatty - taken as a positive outcome.
Visual analogue measure of hunger, satiety, fullness, and prospective food consumption | 4-hours post-intervention
  Satiety Measure recorded on a 100 millimetre scale. Scores closer to 0 millimetres indicate less hunger, less satiety and less fullness - taken as a negative outcome, and less desire for prospective food consumption or consume something sweet, salty, savoury or fatty - taken as a positive outcome.
Visual analogue measure of hunger, satiety, fullness, and prospective food consumption | 6-hours post-intervention
  Satiety Measure recorded on a 100 millimetre scale. Scores closer to 0 millimetres indicate less hunger, less satiety and less fullness - taken as a negative outcome, and less desire for prospective food consumption or consume something sweet, salty, savoury or fatty - taken as a positive outcome.
Visual analogue measure of palatability of the intervention meal | 1-hour post-intervention
  Palatability Measure recorded on a 100 millimetre scale. Scores closer to 0 millimetres indicate good visual appeal, good smell, good taste and good overall palatability - taken as a positive outcome.
Neurotrophic marker | 6-hours post-intervention
  Blood serum levels of BDNF.
Metabolic marker- Glucose | 6-hours post-intervention
  Blood serum levels of glucose
Metabolic marker- Insulin | 6-hours post-intervention
  Blood serum levels of insulin
Metabolic marker- Triglycerides | 6-hours post-intervention
  Blood serum levels of triglycerides (TAG)
Inflammatory marker | 6-hours post-intervention
  Blood serum levels of Interleukin-6 (IL-6)

OTHER OUTCOMES:
Health and Lifestyle Questionnaire | Baseline
  This online survey includes basic demographic questions (eg age, sex, heigh, weight, nationality, disease history and medication use).
Epic-Norfolk Food Frequency Questionnaire (FFQ) | Baseline
  The FFQ is a validated tool for gauging the average habitual dietary intake of micro and macronutrients of an individual in the UK. Data will be processed using the FETA software.
Specialised dietary survey | 6-hours post-intervention on final test day
  Short survey relating to mushroom habitual intake.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Williams, PhD, Principal Investigator — School of Psychology and Clinical Languages, University of Reading
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All personally related collected information, including the paper consent forms, will be kept in locked filing cabinets in the Nutritional Unit of the School of Psychology. The digital health questionnaires used for the purpose of pre-screening participants as well as any digital research data will be stored in the Research Electronic Data Capture (REDCap) database, stored on the University secure network cloud (UREC).
  All relevant study outcomes described in the Ethics Review Application Form (including the demographic and anthropometric data (such as age, sex, BMI, blood pressure) as well as the performance scores of the battery tests assessing cognitive function and mood and the results of the blood tests measuring immunological and metabolic function) will be preserved and made available in anonymised form, so that they can be consulted and re-used by others.

REFERENCES:
- [Background] Ba DM, Gao X, Al-Shaar L, Muscat J, Chinchilli VM, Ssentongo P, Beelman RB, Richie J. Mushroom intake and cognitive performance among US older adults: the National Health and Nutrition Examination Survey, 2011-2014. Br J Nutr. 2022 Dec 14;128(11):2241-2248. doi: 10.1017/S0007114521005195. Epub 2022 Feb 4. PMID 35115063
- [Background] Bingham S, Luben R, Welch A, Low YL, Khaw KT, Wareham N, Day N. Associations between dietary methods and biomarkers, and between fruits and vegetables and risk of ischaemic heart disease, in the EPIC Norfolk Cohort Study. Int J Epidemiol. 2008 Oct;37(5):978-87. doi: 10.1093/ije/dyn111. Epub 2008 Jun 25. PMID 18579574
- [Background] Gregory J, Vengalasetti YV, Bredesen DE, Rao RV. Neuroprotective Herbs for the Management of Alzheimer's Disease. Biomolecules. 2021 Apr 8;11(4):543. doi: 10.3390/biom11040543. PMID 33917843
- [Background] Rahman MA, Abdullah N, Aminudin N. Interpretation of mushroom as a common therapeutic agent for Alzheimer's disease and cardiovascular diseases. Crit Rev Biotechnol. 2016 Dec;36(6):1131-1142. doi: 10.3109/07388551.2015.1100585. Epub 2015 Oct 30. PMID 26514091
- [Background] Kleftaki SA, Simati S, Amerikanou C, Gioxari A, Tzavara C, Zervakis GI, Kalogeropoulos N, Kokkinos A, Kaliora AC. Pleurotus eryngii improves postprandial glycaemia, hunger and fullness perception, and enhances ghrelin suppression in people with metabolically unhealthy obesity. Pharmacol Res. 2022 Jan;175:105979. doi: 10.1016/j.phrs.2021.105979. Epub 2021 Nov 16. PMID 34798266
- [Background] Dicks L, Jakobs L, Sari M, Hambitzer R, Ludwig N, Simon MC, Stehle P, Stoffel-Wagner B, Helfrich HP, Ahlborn J, Ruhl M, Hartmann B, Holst JJ, Ellinger S. Fortifying a meal with oyster mushroom powder beneficially affects postprandial glucagon-like peptide-1, non-esterified free fatty acids and hunger sensation in adults with impaired glucose tolerance: a double-blind randomized controlled crossover trial. Eur J Nutr. 2022 Mar;61(2):687-701. doi: 10.1007/s00394-021-02674-1. Epub 2021 Sep 10. PMID 34505919

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT05594329/Prot_SAP_000.pdf